CLINICAL TRIAL: NCT06626529
Title: Mindful Breaths: A Pilot Randomized Trial on Mindfulness for Young Adult Vaping
Brief Title: Mindful Breaths: Mindfulness for Young Adult Vaping
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Audrey Hai, Assistant Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1480
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Vaping Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness (Experimental): Intervention group participants will practice mindfulness following a ten-minute video of guided mindfulness meditation for craving and addiction.
  Interventions: Behavioral: Guided mindfulness meditation
- Scenery video (Sham Comparator): Control group participants will watch a ten-minute video of calming music and images.
  Interventions: Behavioral: Scenery video

INTERVENTIONS:
Behavioral: Guided mindfulness meditation — Watching a video of a guided mindfulness meditation include paying attention to the breath, promoting natural breathing without force; body scan, directing awareness from the head down to the toes, allowing tension to release in each area. The intervention emphasizes observing sensations without judgment, fostering a state of relaxed awareness.
  Arms: Mindfulness
Behavioral: Scenery video — Watching a ten-minute video of calming music and images
  Arms: Scenery video

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, acceptability, and preliminary efficacy of mindfulness-based interventions (MBI) as a vaping cessation intervention in young adults aged 18-29 who vape nicotine at least 25 days per month and are interested in cutting down or quitting. The main questions it aims to answer are:

* Can mindfulness practice reduce nicotine cravings in young adults?
* Is mindfulness practice an acceptable and feasible intervention for vaping cessation in this population?

Researchers will compare participants in the mindfulness intervention group to a control group that watches a video with calming music and images to see if mindfulness practice has a greater effect on reducing nicotine cravings.

Participants will:

* Complete a baseline survey and craving cue reactivity assessment.
* Engage in a 10-minute guided mindfulness meditation (intervention group) or view calming music and images (control group).
* Rate their cravings and the acceptability, appropriateness, and feasibility of the intervention after the session.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18-29 years old
* Residing in the United States
* Able to read and speak English
* Vape nicotine at least 25 days/month,
* Interested in cutting down or quitting vaping in the next 30 days (rated at least a 5 on a 10-point scale).

Exclusion Criteria:

* Using any nicotine-containing products other than e-cigarettes
* A current or past Diagnostic and Statistical Manual of Mental Disorders (DSM-5) psychiatric diagnosis of severe mental illness
* A current DSM diagnosis of substance use disorders other than tobacco use disorder
* Involved in regular mindful practice
* Undergoing current smoking/vaping cessation treatment (counseling and/or medication)
* Taking any medications that may potentially affect nicotine craving, consumption, or mood within the past 30 days.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction | Within ten minutes after the completion of a single 10-minute guided meditation session
  Satisfaction with the mindfulness intervention will be rated on a scale of 1-5, with a higher score indicating higher satisfaction.
Intervention appeal | Within ten minutes after the completion of a single 10-minute guided meditation session
  Intervention appeal will be rated on a scale of 1-5, with a higher score indicating greater appeal.
Intervention appropriateness | Within ten minutes after the completion of a single 10-minute guided meditation session
  Intervention appropriateness will be rated on a scale of 1-5, with a higher score indicating greater appropriateness.
Intervention feasibility | Within ten minutes after the completion of a single 10-minute guided meditation session
  Intervention feasibility will be rated on a scale of 1-5, with a higher score indicating higher feasibility.
Perceived effectiveness | Within ten minutes after the completion of a single 10-minute guided meditation session
  Perceived intervention effectiveness will be rated on a scale of 1-5, with a higher score indicating greater effectiveness.
Likelihood to continue mindfulness practice | Within ten minutes after the completion of a single 10-minute guided meditation session
  The likelihood of continuing the mindfulness practice will be rated on a scale of 1-5, with a higher score indicating a higher likelihood of continuing the mindfulness practice.

SECONDARY OUTCOMES:
Craving | Within 20 minutes before and after a ten minute guided mindfulness meditation practice.
  Craving for e-cigarettes will be measured with the adapted Visual Analog Craving Scale before and after each cue and the intervention/control to assess their craving intensity. Participants rate craving intensity by selecting a position along a line anchored on the left by "not at all" and on the right by "more than ever."

IPD SHARING:
Plan to Share IPD: No